CLINICAL TRIAL: NCT01419821
Title: Supplemental Vitamin D Administered to One Year Old Vitamin D Deficient Infants Until Age 3 and Its Affect on Growth Rates and Bone Mineral Density Until Age 5
Brief Title: Vitamin D and Its Affect on Growth Rates and Bone Mineral Density Until Age 5
Acronym: VitD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: protocol 5.3
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2011-08

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D; Bone densitometry; Vitamin D supplementation; Growth
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Vit D supplementation (Active Comparator): Group 2-Infants with 25(OH)D below 15ng/ml receiving continued vitamin D supplementation of 800IU (4gtt/d) for one year.
  Interventions: Drug: Vitamin D
- Placebo group (Placebo Comparator): Group 3- Infants with 25(OH)D below 15ng/ml those receiving the placebo.
  Interventions: Other: Placebo (for Vitamin D)
- Normal group (No Intervention): Group 1- infants with 25(OH)D above 15ng/ml (normal levels) will receive no intervention.

INTERVENTIONS:
Drug: Vitamin D — 800IU (4gtt/d) once a day for 2 years once a day.
  Other Names: TipTipot Vitamin D 200IU/gtt
  Arms: Vit D supplementation
Other: Placebo (for Vitamin D) — 4gtt/d for the placebo for two years.
  Arms: Placebo group

SUMMARY:
Abstract Background: Vitamin D affects a wide variety of functions in the body including regulation of calcium, phosphorus, and bone metabolism. Israeli studies have documented a high prevalence of Vitamin D deficiency in Israeli infants in general, which was more severe in infants from Ultra-Orthodox Jewish families. Modest dress requirements in this population drastically reduce sun exposure, known to encourage production of Vitamin D. Countless research has analyzed preterm as well as term neonates born to mothers with vitamin D deficiency, with regard to weight, height, and bone mineral density at birth. However, there is a paucity of information about healthy infants' vitamin D levels and its' correlation to these parameters during the first few years of life. Objectives: The purpose of the proposed study is to measure and correlate levels of 25(OH)D and bone mineral density towards the end of the first year of life with growth rates and bone mineral density in the same children at the ages of 2, 3 and 5 years. Patients and Methods: The study will be performed in the Ultra-Orthodox Jewish community of Beitar Illit. 25(OH)D levels will be taken between 9-12 months of age (when routine blood tests are normally drawn for these infants) and bone mineral density will be measured using Quantitative Ultrasound. Infants will be divided into 2 groups: those with those with normal 25(OH)D levels (>15ng/ml), and those with 25(OH)D deficiency (<15ng/ml). Group 1- normal levels will receive no intervention. Infants with 25(OH)D below 15ng/ml will be randomly assigned into one of two groups; Group 2-those receiving continued vitamin D supplementation of 800 international units(IU) (4gtt/d) for one year, or Group 3- those receiving the placebo. Height, weight, and head circumference growth curves will be recorded every two months until 2 years of age. Quantitative ultrasound, growth charts and blood tests including 25(OH)D, serum calcium and phosphate levels, Parathyroid hormone (PTH), and alkaline phosphatase, taken at approximately 9-12 months will be repeated at 2 years of age. At that time children from Group 1 (no supplementation) will be divided into three: Group 1a- normal 25(OH)D levels will continue with no intervention, Group 1b <15ng/ml will begin receiving vitamin D 4gtt/d, Group 1c <15ng/ml will receive a placebo until age three. Groups 2 and 3 will continue their previous treatment until age three. All aforementioned tests will be repeated at age 3, when treatment will stop, and the same tests will be repeated at age 5.

ELIGIBILITY:
Inclusion Criteria:

Infants between 9-12 months old in Tipat Chalav and Kupat Holim Clalit in Beitar Illit undergoing a blood draw for CBC at one year of age.

Exclusion Criteria:

Parents that refuse to participate in this study, infants with any diagnosed chronic disease, and preterm infants less than 34 weeks.

Ages: 9 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Height at the age of 3 years | 3 years after the recruitment begins

SECONDARY OUTCOMES:
Bone densitometry by ultrasound | 3 years after recruitment begins

CONTACTS AND LOCATIONS:
Overall Officials: Avigdor Hevroni, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Clalit Health services, Beitar Elit, Israel

REFERENCES:
- [Background] Greer FR. Issues in establishing vitamin D recommendations for infants and children. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1759S-62S. doi: 10.1093/ajcn/80.6.1759S. PMID 15585801